CLINICAL TRIAL: NCT05087355
Title: Health Status Prior and Post Infection With Influenza or COVID 19: a Population Based Retrospective Analysis of 2016-2021
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Landesklinikum Sankt Polten (Other); Sicknessfund Burgenland (BGKK) (Unknown); A.ö. Krankenhaus St. Josef Braunau GmbH (Other)
Responsible Party: Principal Investigator, Hendrik Jan Ankersmit, Principal Investigator/Univ. Prof. , MD, MBA, Medical University of Vienna
Other Study IDs: AUTCOV-INFLU-STUDY
Record Dates: First submitted 2021-10-19; First posted 2021-10-21 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Covid 19; Influenza
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Influenza
  Interventions: Diagnostic Test: PCR or antigen test for Covid 19 or Inluenza
- Covid 19
  Interventions: Diagnostic Test: PCR or antigen test for Covid 19 or Inluenza
- Control group: hospitalisation due to other disease (not influenza or Covid 19)
  Interventions: Diagnostic Test: PCR or antigen test for Covid 19 or Inluenza

INTERVENTIONS:
Diagnostic Test: PCR or antigen test for Covid 19 or Inluenza — PCR or antigen test for Covid 19 or Inluenza

SUMMARY:
The overall project aim is to study outcomes after COVID-19 and influenza hospitalisation from 2016 - 2021 by retrieving data from the main social security carriers in Austria for the years 2010-2018

ELIGIBILITY:
Inclusion Criteria:

* Patients with SARS
* Patients with Covid-19
* Patients after Covid-19
* Patients with influenza

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with or after Covid-19 or influenza between 2016-2021 in Austria will be included in this study
Sampling Method: Non-Probability Sample
Enrollment: 440000 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Overall Mortality | 5 years
  Overall mortality after influenza or covid-19
age distribution | 5 years
  age distribution in patients with influenza or covid-19
risk profile | 5 years
  risk profile (e.g. prior diseases, medication) in patients who died due to influenza or covid-19
newly diagnosed diseases | 5 years
  newly diagnosed diseases after influenza or covid-19
newly prescribed medication | 5 years
  newly prescribed medication after influenza or covid-19
duration of hospitalisation or unemployability | 5 years
  duration of hospitalisation or unemployability after influenza or covid-19